CLINICAL TRIAL: NCT06736080
Title: A Phase I/II Open Label Non Randomized Study, Monocentric, Single Arm, Evaluating Safety and Efficacy of Gene Therapy of FHL 3 Caused by Mutations in the Human UNC13D Gene by Transplantation of a Single Dose of Autologous CD34+ Cells Transduced Ex Vivo with the UNC13D LV Vector Expressing the UNC13D CDNA
Brief Title: Safety and Efficacy of Gene Therapy of FHL Type 3 Caused by Mutations in the Human UNC13D Gene by Transplantation of a Single Dose of Autologous CD34+ Cells Transduced Ex Vivo with the UNC13D LV Vector Expressing the UNC13D CDNA
Acronym: MUNC13-4
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP240201; 2023-507334-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Familial Hemophagocytic Lymphohistiocytosis Type 3 (FHL 3)
Keywords: Familial Hemophagocytic Lymphohistiocytosis type 3 (FHL 3); Munc13.4; Gene Therapy; Lentiviral Vector

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MUNC (Experimental)
  Interventions: Drug: MUNC-CD34; Drug: MUNC-T3

INTERVENTIONS:
Drug: MUNC-CD34 — * Dosage: ≥ 2 x10e6 CD34/kg after thawing, dose limit: 20x10e6 CD34+ cells/kg
  * Route of administration: intravenous, on D0
Drug: MUNC-T3 — * Dosage: [1.10e4; 5.10e6] T-CD3+/kg after thawing,
  * Route of administration: intravenous, on D14 post-GT +/- D28 In case of persistent circulating T-cell after the HLH remission at inclusion, the MUNC-CD34 will be completed by MUNC-T3 infusion

SUMMARY:
The investigators propose to replace HLA- partially compatible allogeneic Hematopoietic Stem Cell Transplantation (HSCT) for FHL type 3 patients, with autologous transplantation of immunoselected gene-modified CD34+ cells, combined with transduced autologous T-cell each time this is possible and also to propose this alternative treatment as salvage in case of failure of a previous allogeneic HSCT. This approach should avoid the severe immunological complications (failure to engraft, acute or chronic graft versus host disease (GVHD)) and conditioning toxicities such as severe Veno-Occlusive Disease (VOD). As the clinical manifestations of FHL type 3 patients are triggered by opportunistic viral infections (often EBV) and can be poorly controlled or only transiently controlled by the available drugs , providing the patient after the conditioning with immediately functional autologous cytotoxic T-cells could be key to maintain the control of the viral infection and hopefully its eradication awaiting for the hematopoietic reconstitution . This procedure should avoid any reactivation of the viral infection and thus improving the patients' overall survival and event-free survival while clearing the ongoing triggering infections.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged from 3 months up to 17 years old.
2. Patient with a FHL caused by mutation of the UNC13D gene.
3. Complete remission is defined by the normalization of clinical and laboratory parameters:

   1. Resolution of fever
   2. Resolution of splenomegaly or reduced and isolated splenomegaly.
   3. Improvement of cytopenia: absolute neutrophil count > 500/µl AND platelets cout > 100 000/ µl (unsupported by transfusion)
   4. Normalization of serum fibrinogen level (Fibrinogen ≥1.5g/l)
   5. Resolution of hyperferritinemia (Ferritin level < 2000µg/l)
   6. Normalization of T-cell activation
4. Patient eligible for an allogeneic HSCT in absence of an HLA geno-identical donor (at diagnostic or 6 months after failure of a previous HSCT (rejection or loss of the graft))
5. Parental, guardian's patient signed informed consent.
6. For patients of childbearing age : willing to use an effective method of contraception* during the trial and for at least 12 months post-infusion
7. Affiliation to Social Security

Exclusion Criteria:

1. Active CNS encephalitis related to HLH
2. Existence of a matched -sibling donor
3. Unwillingness to return for follow-up during the 2 years study and lifelong for off study review.
4. HIV-1 or 2 or HTLV1 infections.
5. Patient on AME (state medical aid) (unless exemption from affiliation)
6. Pregnancy or breast feeding in a post-partum female
7. Diagnosis of significant psychiatric disorder of the subject that could seriously impeded the ability to participate in the study
8. Known allergies, hypersensitivity, or intolerance to any of busulfan, fludarabine, rituximab, G-CSF, plerixafor or excipients, or similar compounds
9. Unable to tolerate general anesthesia and/or apheresis
10. Participation in another clinical study with an investigational drug within 30 days of inclusion.
11. Uncontrolled HLH manifestation

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Transplantation Related Mortality (TRM) | up to 6 months post treatment
Frequency and severity of clinical AEs and laboratory parameters | throughout the whole period of the research, up to 60 months
  Adverse event will be measured using CTCAE
Incidence of clinically detectable malignancy and/or abnormal clonal dominance assessed as related to study treatment | At 12 months post treatment
  Bone marrow analysis and VISA
Detection of Replication -Competent Lentivirus (RCL) | at 3, 6 and 12 months post treatment, then yearly up to 60 months

SECONDARY OUTCOMES:
Neutrophil and platelet recovery | throughout the whole period of the research, up to 60 months
  ANC> 500/µl, Platelets > 20.000/µl on two consecutive days without transfusion
Quantification of the transgene copy number (VCN) on drug substance at time of cryopreservation, on PBMC, sorted T-CD3+ and sorted NK cells | at 1, 2, 3, 6, 9, 12, 18 and 24 months post treatment
Quantification of the UNC13D RNA on PBMC | at 1, 2, 3, 6, 9, 12, 18 and 24 post treatment
  by Q-PCR
Quantification of Munc13.4 protein level in the drug substance and on peripheral blood mononuclear cells and on sorted CD3+ and CD56+ cells in function of their number | at 6, 12 and 24 months post treatment
  by western blot
Determination of the total number of T-cells and distribution of different subpopulations | at 1, 2, 3, 6, 12, 18 and 24 months post treatment
  Naïve and memory CD4+ and CD8+ T cells will be evaluated using CCR7/CD45RA/RO markers, and the quantification of activation marker will be performed by the expression of DR+. by flow cytometry
Correction of degranulation function in T-CD3 | at 6 months and 24 months post treatment
Integration site analyse study | at 24 months post treatment
Needs of PICU support | up to 24 months post treatment
Endothelial complications | up to 24 months post treatment
Infectious diseases | up to 24 months post treatment
Estimate of the cost of the complete procedure, from mobilisation to transplant | up to 24 months post treatment
stimate of the 24 months total cost | up to 24 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien DIANA, MD, PhD, Study Director — Assitance publique - Hôpitaux de Paris; Chantal LAGRESLE, PHD, Study Chair — Inserm Institut Imagine
Locations (1):
- Hôpital Necker Enfant Malades, Paris, France